CLINICAL TRIAL: NCT02099513
Title: The Mobile Health Platform - Development and Feasibility Evaluation
Brief Title: The Mobile Health Platform
Acronym: mHealth
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: Pro00048816
Record Dates: First submitted 2014-03-26; First posted 2014-03-31 (Estimated); Last update posted 2017-02-23 (Actual); Status verified 2014-10

CONDITIONS: Obesity; Hypertension; Diabetes
Keywords: Mobile Technology; Chronic illness; Wireless blood pressure device; Wireless scale; Pedometer
MeSH Terms: conditions — Obesity; Hypertension; Diabetes Mellitus; Chronic Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: The Mobile Health Platform
  Other Names: mHealth

SUMMARY:
This study develops and pilots the initial interface of our mobile health platform that will allow for intra-individual tailoring and personalization of health interventions. This will allow for just-in-time interventions that adapt both the content and timing, not just initially, but also over time based upon prior outcome data, responses to an intervention, current environmental and social context, activity level, location, time, and an individual's psychophysiological state.1,2

Aim 1: To develop the initial interface of the mobile health platform that will allow patients to report and receive data representing multiple health domains including blood pressure, pO2 (pulse oximeter), values, weight, physical activity, calories burned, sleep, and self-report survey measures such as pain and fatigue.

Aim 2: To assess feasibility of the mobile health platform to receive and deliver data representing multiple health domains over 1 month through a single-case study design (N=6).3 Aim 3: To develop an algorithm using the diet data collected in Aim 1 that will facilitate adaptive work by providing patients with automated real time feedback on their progress.

Aim 4: To develop an algorithm using the diet data collected in Aim 1 that will that will facilitate adaptive approaches by alerting clinicians on the progress of their patients.

DETAILED DESCRIPTION:
At baseline we will collect demographic variables and acceptance and use of technology from surveys, and biological variables including blood pressure, weight, and blood glucose from electronic medical records. Over a period of 1 month, participants will be asked to track and collect daily data on weight using the iHealth wireless scale. Participants will also collect blood pressure (BP), pO2, and pulse using the iHealth blood pressure device. Physical activity and sleep activity will be measured using the fitbit device. Participants will receive evidence-based daily nutrition and exercise weight loss messages via text messages.

Following the one-month observation participants will be asked to complete a follow-up survey on acceptance and use of technology and to undergo a post-formative semi-structure telephone interview to discuss their perception of the usefulness and attitudes toward the platform, technical difficulties and barriers, and recommendations for future development.

ELIGIBILITY:
Inclusion Criteria:

* Patient of Picket primary care clinic
* All subjects will provide written informed consent.
* Three participants who have multiple chronic illnesses.
* Chronic illnesses of obesity (BMI>29)
* Chronic hypertension (SBP>140)
* Three healthy participants who do not have any chronic illnesses.
* Own a smartphone with a data and text messaging plan.
* Have Wifi available in the home.

Exclusion Criteria:

* No internet/Wifi available in the home.
* No Smartphone

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2014-03; Primary Completion 2014-10 (Actual); Study Completion 2014-10 (Actual)

PRIMARY OUTCOMES:
Change in the Acceptance and use of technology survey | Baseline, up to 1 Month
  Subject will take survey at Baseline, and the 1 month mark.
Perception of perceived usefulness, attitudes, and experiences | 1 month
  Questions will be asked in the interviews regarding perceived usefulness, attitudes, and experiences of the mHealth applications. The results will be divided into three main categories of positive, negative, and neutral perceptions.

CONTACTS AND LOCATIONS:
Overall Officials: Ryan J. Shaw, RN, Phd, Principal Investigator — Duke University
Locations (1):
- Duke University Medical Center, Pickens Primary Care Clinic, Durham, North Carolina, United States